CLINICAL TRIAL: NCT02201056
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability and Pharmacokinetic Study of Escalating Single Doses of TAK-935 in Healthy Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of Escalating Single Doses of TAK-935
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-935_101; U111-1155-6022 (Registry Identifier: WHO)
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Results first posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort 1: TAK-935 15 mg (Experimental): TAK-935 15 mg solution, orally, once, on Day 1.
  Interventions: Drug: TAK-935
- Cohort 2: TAK-935 50 mg (Experimental): TAK-935 50 mg solution, orally, once, on Day 1.
  Interventions: Drug: TAK-935
- Cohort 3: TAK-935 200 mg (Experimental): TAK-935 200 mg solution, orally, once, on Day 1.
  Interventions: Drug: TAK-935
- Cohort 4: TAK-935 600 mg (Experimental): TAK-935 600 mg solution, orally, once, on Day 1.
  Interventions: Drug: TAK-935
- Cohort 5: TAK-935 900 mg (Experimental): TAK-935 900 mg solution, orally, once, on Day 1.
  Interventions: Drug: TAK-935
- Cohort 6: TAK-935 1350 mg (Experimental): TAK-935 1350 mg solution, orally, once, on Day 1.
  Interventions: Drug: TAK-935
- Cohorts 1-6: Placebo (Placebo Comparator): TAK-935 placebo-matching solution, orally, once, on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-935 — TAK-935 oral solution
  Arms: Cohort 1: TAK-935 15 mg; Cohort 2: TAK-935 50 mg; Cohort 3: TAK-935 200 mg; Cohort 4: TAK-935 600 mg; Cohort 5: TAK-935 900 mg; Cohort 6: TAK-935 1350 mg
Drug: Placebo — TAK-935 placebo-matching oral solution
  Arms: Cohorts 1-6: Placebo

SUMMARY:
The purpose of this study is to characterize the safety and tolerability profile of TAK-935 in healthy participants when administered as a single dose of oral solution at escalating dose levels.

DETAILED DESCRIPTION:
The drug being tested in this study is TAK-935. TAK-935 is being tested to find a safe and well-tolerated dose and to assess how TAK-935 is processed by the body. This study will look at side effects and lab results in people who take TAK-935 and is designed as a randomized dose-rising study.

The study will consist of 6 Cohorts with 8 participants in each Cohort. In each Cohort, 6 participants will receive a single dose of TAK-935 and 2 participants will receive placebo after a 10-hour fast. The starting dose will be 15 mg followed by planned doses of 50, 200, 600, 900 and not to exceed 1350 mg in subsequent cohorts.

This single-center trial will be conducted in the United States. The overall time to participate in this study is up to 51 days. Participants will make 2 visits to the clinic, including one 7-day period of confinement to the clinic. All participants will be contacted by telephone 14 days after the dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female adult who is 19 to 55 years of age inclusive at the time of informed consent.
2. Weighs at least 45 kg and has a body mass index (BMI) between 18.0 and 30.0 kg/m^2, inclusive at the Screening Visit.

Exclusion Criteria:

1. Has uncontrolled, clinically significant neurological (including seizure disorders), cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urological, immunologic, endocrine disease, or psychiatric disorder, or other abnormality.
2. Has a known hypersensitivity to any component of the formulation of TAK-935.
3. There is any finding in the participant's medical history, significant results from physical examination, or safety laboratory tests.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Lincoln, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 09 July 2014 to 30 July 2015.
Pre-assignment Details: Healthy Volunteers were enrolled in 1 of 7 treatment groups, once a day placebo, TAK 935 15 mg, 50 mg, 200 mg, 600 mg, 900 mg or 1350 mg.
Period: Overall Study
Arm/Group | Cohorts 1-6: Placebo | Cohort 1: TAK-935 15 mg | Cohort 2: TAK-935 50 mg | Cohort 3: TAK-935 200 mg | Cohort 4: TAK-935 600 mg | Cohort 5: TAK-935 900 mg | Cohort 6: TAK-935 1350 mg
Started | 12 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 12 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety set which included all participants who were enrolled and received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohorts 1-6: Placebo | Cohort 1: TAK-935 15 mg | Cohort 2: TAK-935 50 mg | Cohort 3: TAK-935 200 mg | Cohort 4: TAK-935 600 mg | Cohort 5: TAK-935 900 mg | Cohort 6: TAK-935 1350 mg | Total
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (10.41) | 34.2 (8.21) | 34.3 (10.93) | 29.8 (6.74) | 35.3 (13.31) | 30.5 (10.33) | 32.8 (12.97) | 33.6 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 0 | 0 | 2 | 6 | 6 | 22
  Male | 7 | 3 | 6 | 6 | 4 | 0 | 0 | 26
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 2 | 0 | 1 | 0 | 2 | 2 | 1 | 8
  White | 10 | 6 | 5 | 6 | 3 | 4 | 5 | 39
  Multiracial | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 4
  Non-Hispanic or Latino | 11 | 4 | 5 | 6 | 6 | 6 | 6 | 44
Region of Enrollment [Number; unit: participants]
  United States | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Height [Mean (Standard Deviation); unit: cm] | 170.8 (5.99) | 165.0 (11.52) | 175.0 (5.59) | 178.7 (7.31) | 173.5 (8.89) | 161.5 (2.88) | 165.5 (2.59) | 170.1 (8.43)
Weight [Mean (Standard Deviation); unit: kg] | 70.23 (10.478) | 68.88 (19.873) | 78.25 (13.623) | 80.18 (12.039) | 76.85 (9.465) | 70.10 (6.214) | 69.28 (10.981) | 73.00 (12.178)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.00 (2.532) | 24.86 (4.073) | 25.44 (3.361) | 25.05 (3.039) | 25.51 (2.539) | 26.88 (2.313) | 25.34 (4.251) | 25.13 (3.064)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience at Least One Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug and within 30 days after the last dose of study drug.
Time Frame: Day 1 to Day 30
Population: Safety set included all participants who were enrolled and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohorts 1-6: Placebo | Cohort 1: TAK-935 15 mg | Cohort 2: TAK-935 50 mg | Cohort 3: TAK-935 200 mg | Cohort 4: TAK-935 600 mg | Cohort 5: TAK-935 900 mg | Cohort 6: TAK-935 1350 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants | 41.7 | 33.3 | 16.7 | 33.3 | 83.3 | 33.3 | 33.3

2. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria, for Safety Laboratory Tests at Least Once Post-dose
Description: The percentage of participants with any markedly abnormal standard safety laboratory values (hematology, serum chemistries, and urinalysis) collected during the treatment period.
Time Frame: Day 1 to Day 14
Population: Safety set included all participants who were enrolled and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohorts 1-6: Placebo | Cohort 1: TAK-935 15 mg | Cohort 2: TAK-935 50 mg | Cohort 3: TAK-935 200 mg | Cohort 4: TAK-935 600 mg | Cohort 5: TAK-935 900 mg | Cohort 6: TAK-935 1350 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants | 16.7 | 0 | 0 | 0 | 0 | 16.7 | 0

3. Primary Outcome: Percentage of Participants Who Meet Markedly Abnormal Criteria, for Vital Sign Measurements at Least Once Post-dose
Description: The percentage of participants with any markedly abnormal vital signs (oral temperature, respiration rate, pulse, and blood pressure) collected during the treatment period.
Time Frame: Day 1 to Day 14
Population: Safety set included all participants who were enrolled and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohorts 1-6: Placebo | Cohort 1: TAK-935 15 mg | Cohort 2: TAK-935 50 mg | Cohort 3: TAK-935 200 mg | Cohort 4: TAK-935 600 mg | Cohort 5: TAK-935 900 mg | Cohort 6: TAK-935 1350 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants | 75.0 | 100 | 66.7 | 66.7 | 66.7 | 66.7 | 66.7

4. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria, for Electrocardiogram (ECG) Measurements at Least Once Post-dose
Description: The percentage of participants with any markedly abnormal criteria for standard 12-lead ECG measured collected during the treatment period.
Time Frame: Day 1 to Day 14
Population: Safety set included all participants who were enrolled and received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohorts 1-6: Placebo | Cohort 1: TAK-935 15 mg | Cohort 2: TAK-935 50 mg | Cohort 3: TAK-935 200 mg | Cohort 4: TAK-935 600 mg | Cohort 5: TAK-935 900 mg | Cohort 6: TAK-935 1350 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants | 25.0 | 66.7 | 83.3 | 50.0 | 16.7 | 33.3 | 33.3

5. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-935
Time Frame: Multiple time-points (Up to 96 hours) post-dose
Population: Pharmacokinetic (PK) set included all participants in the safety set who had at least 1 measurable plasma or urine concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: TAK-935 15 mg | Cohort 2: TAK-935 50 mg | Cohort 3: TAK-935 200 mg | Cohort 4: TAK-935 600 mg | Cohort 5: TAK-935 900 mg | Cohort 6: TAK-935 1350 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 43.533 (41.2350) | 210.150 (153.0463) | 571.167 (257.8002) | 4551.667 (2573.5067) | 5080.000 (1801.9323) | 7953.333 (2151.3035)

6. Secondary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-935
Time Frame: Multiple time-points (Up to 96 hours) post-dose
Population: PK set included all participants in the safety set who had at least 1 measurable plasma or urine concentration.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1: TAK-935 15 mg | Cohort 2: TAK-935 50 mg | Cohort 3: TAK-935 200 mg | Cohort 4: TAK-935 600 mg | Cohort 5: TAK-935 900 mg | Cohort 6: TAK-935 1350 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 33.323 (28.9569) | 168.736 (88.3702) | 562.660 (196.6517) | 5791.561 (3427.9888) | 7619.088 (1928.2091) | 13501.049 (5778.0847)

7. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity of TAK-935
Time Frame: Multiple time-points (Up to 96 hours) post-dose
Population: PK set included all participants in the safety set who had at least 1 measurable plasma or urine concentration.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cohort 1: TAK-935 15 mg | Cohort 2: TAK-935 50 mg | Cohort 3: TAK-935 200 mg | Cohort 4: TAK-935 600 mg | Cohort 5: TAK-935 900 mg | Cohort 6: TAK-935 1350 mg
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 6 | 6
ng*hr/mL | 23.290 (6.7061) | 172.430 (107.0799) | 621.369 (240.5953) | 5809.066 (3427.5393) | 7660.961 (1962.0905) | 13541.772 (5763.4722)

ADVERSE EVENTS:
Time Frame: 30 Days
Description: At each visit the investigator had to document any occurrence of adverse events, including and abnormal clinically significant abnormal laboratory values or ECG findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment and/or intensity.
Arm/Group | Cohorts 1-6: Placebo | Cohort 1: TAK-935 15 mg | Cohort 2: TAK-935 50 mg | Cohort 3: TAK-935 200 mg | Cohort 4: TAK-935 600 mg | Cohort 5: TAK-935 900 mg | Cohort 6: TAK-935 1350 mg
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/12 | 2/6 | 1/6 | 2/6 | 5/6 | 2/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohorts 1-6: Placebo (N=12) | Cohort 1: TAK-935 15 mg (N=6) | Cohort 2: TAK-935 50 mg (N=6) | Cohort 3: TAK-935 200 mg (N=6) | Cohort 4: TAK-935 600 mg (N=6) | Cohort 5: TAK-935 900 mg (N=6) | Cohort 6: TAK-935 1350 mg (N=6)
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Application site dermatitis (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Application site erosion (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Application site erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Application site pruritus (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 2 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.